CLINICAL TRIAL: NCT04448093
Title: Relationship Between Quality of Life, Self-image and Oral Health in Patients Undergoing Hemodialysis: A Comparative Study.
Brief Title: Relationship Between Quality of Life, Self-image and Oral Health in Patients Undergoing Hemodialysis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Olga Flecha, Principal Investigator, Federal University of São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hemodialysis
Record Dates: First submitted 2020-03-09; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Patients Undergoing Hemodialysis
Keywords: Quality of life; Dentistry; Renal dialysis; Epidemiology; Self-image
MeSH Terms: interventions — Dental Care

STUDY DESIGN:
Intervention Model Description: Intervention group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Treated group (53) that answered quality of life questionnaires before, after and with 45 days of treatment.
  Interventions: Procedure: dental treatment
- Group control (No Intervention): Untreated group (68) that answered quality of life questionnaires before, after and with 45 days of treatment.

INTERVENTIONS:
Procedure: dental treatment — Dental treatment of adequacy of oral environment and assessment of quality of life and self-esteem through questionnaires comparing a group that received treatment with another that did not.
  Arms: Treatment group

SUMMARY:
The objective of this work will be to conduct a controlled clinical trial to assess whether the dental treatment of adequacy of the oral environment is capable of generating improvement in the quality of life and self-esteem, comparing the results of patients on hemodialysis who received treatment with others who did not receive treatment .

DETAILED DESCRIPTION:
After selecting the sample, patients will undergo an oral examination performed by a dental surgeon, in which they will be evaluated for the presence of lesions in the oral mucosa, periodontal conditions through simplified periodontal record - PSR, oral hygiene index, caries and lack of teeth - DMFT, if they need treatment and the situation of the prosthesis, if they use them, the data being recorded in a specific medical record. Subsequently, intervention will be performed in the group that received the treatment (intervention group). The treatment will consist of the adequacy of the oral environment in patients with teeth and evaluation of the mucosa and prostheses for edentulous patients.

The service will take place at the UFVJM Surgery and Periodontics Clinic, on previously scheduled days and times. About 5 to 10 days before treatment, patients answered questionnaires about socioeconomic characterization, self-esteem and quality of life. The therapeutic protocol followed during the service will be the one proposed by Quirynen (1995) [22], in which the debridement of the entire mouth is recommended in a single 45-minute session. After removing the supra and subgingival biofilm, the patient will be instructed to use mouthwashes with 15 ml of 0.12% chlorhexidine gluconate, for one minute, twice a day, thirty minutes after brushing, for seven days. In this phase, emergency extractions, restoration of restorations and cavity closure with glass ionomer cement and resins in the anterior teeth will also be performed, in order to adapt the oral environment in minimal interventions, considering the patient's systemic state.

All patients who have at least 1 tooth, healthy or not, will be considered dentate. Toothless patients will receive guidance on oral hygiene and prostheses, if used, and will also use mouthwash with 0.12% chlorhexidine gluconate for the same period. Group participants who were not submitted to the intervention (control group), received the same initial assessment and answered the same questionnaires, but will not be treated at that time. After 45 days from the end of the dental treatment, everyone will be reassessed, went through oral hygiene instructions again and answered the questionnaires, the questions being directed to the patient's perception in the last 45 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years
* submitted to hemodialysis
* agreed to participate voluntarily by invitation and sign an informed consent form

Exclusion Criteria:

* severe anemia
* uncontrolled systolic and diastolic blood pressure or greater than 180/110 mmHg
* unstable angina, complex ventricular arrhythmias, severe metabolic disease
* acute myocardial infarction less than a month
* acute conditions, aortic aneurysm, severe aortic stenosis or respiratory impairment
* neurological and / or musculoskeletal that contraindicate treatment

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2015-08-29 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Dental treatment | 6 years
  Comparison of quality of life and self-esteem results of patients who underwent dental treatment with others who did not.

CONTACTS AND LOCATIONS:
Locations (1):
- Periodontics Clinic, Department of Dentistry, Diamantina, Minas Gerais, Brazil